CLINICAL TRIAL: NCT07091370
Title: A Multicenter, Open-label, Single-arm Phase I Clinical Trial on the Safety and Tolerability of Inaticabtagene Autoleucel Injection in the Treatment of Autoimmune Hemolytic Anemia That Has Failed at Least Three Lines of Treatment
Brief Title: Inaticabtagene Autoleucel Injection in the Treatment of Autoimmune Hemolytic Anemia After Three or More Lines of Therapy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY001106
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: AIHA - Cold Autoimmune Hemolytic Anemia
Keywords: AIHA; CarT
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Inaticabtagene Autoleucel Injection (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, Inaticabtagene Autoleucel Injection.
  Interventions: Drug: Inaticabtagene Autoleucel Injection

INTERVENTIONS:
Drug: Inaticabtagene Autoleucel Injection — The dose was incremented according to the "3+3" principle, and the three dose levels A, B and C were given in sequence at one time, which were respectively:
  A-1 dose group: 0.25×10^6 CAR-T live cells /kg body weight
  Group A (initial dose) : 0.5×10^6 CAR-T live cells /kg body weight
  Group B: 1.0×10^6 CAR-T live cells /kg body weight
  Group C: 1.5×10^6 CAR-T live cells /kg body weight

SUMMARY:
This is a multicenter, open-label, single-arm Phase I clinical trial to evaluate the safety and tolerability of Inaticabtagene Autoleucel Injection treatment in autoimmune hemolytic anemia that has failed at least three lines of treatment.

DETAILED DESCRIPTION:
This study will be conducted in Chinese hospitals and to include 6 to 12 subjects with autoimmune hemolytic anemia .

The main purpose of the study is to evaluate the safety and tolerability of Inaticabtagene Autoleucel Injection in the treatment of autoimmune hemolytic anemia that has failed at least three lines of treatment, and determine the recommended phase II dose (RP2D) of Inaticabtagene Autoleucel Injection in subjects with autoimmune hemolytic anemia who have failed at least three lines of treatment.

The Secondary purpose of the study is to evaluate the efficacy of Inaticabtagene Autoleucel Injection in the treatment of autoimmune hemolytic anemia that has failed at least three lines of treatment and to evaluate the pharmacokinetic (PK) characteristics, pharmacodynamic (PD) characteristics and immunogenicity in the treated patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-75 years (including 18 and 75 years), regardless of gender.
2. Clinically diagnosed with AIHA or Evans, with hemoglobin lower than 100g/L and symptoms related to anemia according to the diagnostic criteria of the "Diagnosis and Treatment Guidelines for Autoimmune Hemolytic Anemia in Chinese Adults (2023 Edition)" and the "Chinese Expert Consensus on the Diagnosis and Treatment of Evans Syndrome (2024 Edition)". And meet the diagnostic criteria of failure in at least three lines of treatment as follows:

   Patients diagnosed with warm resistance type AIHA (wAIHA)/mixed AIHA (mAIHA) /Evans syndrome, the following conditions must be met: first-line glucocorticoid treatment failed, second-line rituximab treatment failed and failure of third-line treatment measures (including any one or more of splenectomy, cyclosporine, cyclophosphamide, azathioprine, mycophenolate mofetil, fludarabine, bortezomib, etc.) Patients diagnosed with cold-resistant type AIHA (cAIHA), that is, cold agglutinin disease (CAD), the following conditions must be met: first-line rituximab treatment failed, second-line rituximab ± bendamustine/fludarabine failed and failure of third-line treatment measures (including any one or more of bortezomib, cyclosporine, cyclophosphamide, mycophenolate mofetil, azathioprine, etc.)
3. Women of childbearing potential must have a negative blood pregnancy test during the screening period. Any male and female patients of childbearing potential must agree to use an effective method of contraception throughout the study and for at least 2 year following infusion of CAR-T cells. Childbearing potential is biologically capable of bearing a living baby and sexually active. Female patients who were not of childbearing potential (ie, met at least 1 of the following criteria):

   Hysterectomy or oophorectomy, or medically confirmed ovarian failure, or medically confirmed postmenopausal (cessation of menses for at least 12 consecutive months in the absence of pathological or physiological causes).
4. Adequate organ function according to the following criteria:

   Aspartate aminotransferase (AST) ≤ 3 times of upper limit of normal (ULN); Alanine aminotransferase (ALT) ≤ 3 times ULN; Serum creatinine ≤ 1.5 times ULN, or creatinine clearance ≥ 60 mL/min (Cockcroft and Gault formula); International normalized ratio (INR) ≤ 1.5 times ULN, and activated partial thromboplastin time (APTT) ≤ 1.5 times the ULN; Must have minimal pulmonary reserve and oxygen saturation > 93% in a nonoxygenated state;
5. The Eastern Cancer Consortium (ECOG) performance status score is 0-2.

Exclusion Criteria:

1. Previously diagnosed proliferative tumors of the lymphatic system;
2. Secondary AIHA caused by drugs or infections;
3. Pregnancy or breastfeeding;
4. Previously undergone organ or hematopoietic stem cell transplantation;
5. A history of new thrombosis or organ infarction within 6 months prior to screening;
6. The active stage diagnosed as a connective tissue disease;
7. Suffering from hereditary hemolytic diseases or other acquired hemolytic diseases;
8. Combined with active infections (such as sepsis, bacteremia, mycosis, uncontrolled pulmonary infection and active tuberculosis, etc.);
9. Positive for hepatitis B surface antigen (HBsAg) and/or hepatitis Be antigen (HBeAg); Hepatitis Be antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) are positive, and the HBV-DNA copy number is greater than the measurable lower limit; Positive for hepatitis C (HCV) antibody; Positive for human immunodeficiency virus (HIV) antibody; Those with positive syphilis (TP) test;
10. Major surgery that was assessed as unsuitable by the investigators within 4 weeks before screening;
11. Patients with concurrent active malignancy within the past five years, those with a history of malignancy but cuired are eligible.
12. The patient's heart meets any of the following conditions:

    * Left ventricular ejection fraction (LVEF) ≤45%;
    * New York Heart Association (NYHA) grade III or IV congestive heart failure or active heart disease;
    * Severe arrhythmias requiring treatment (excluding atrial fibrillation and paroxysmal supraventricular tachycardia);
    * The QTcB interval was ≥450ms for males and ≥470ms for females (QTcB=QT/ R1/2);
    * Had myocardial infarction, bypass surgery or stent surgery within 6 months before the study;
    * Other heart diseases judged by the researchers as unsuitable for inclusion in the group;
13. Have received live vaccines within 6 weeks before screening.
14. Patients participating in any other interventional clinical study or receiving treatment of an active investigational drug within 3 months or 5 half-lives for launched drugs prior to Inaticabtagene Autoleucel Injection infusion.
15. Patients with a history of epilepsy, cerebral ischemia/hemorrhage, cerebellar diseases, or other active central nervous system disorders;
16. Patients with hypersensitivity reactions to the components of Inaticabtagene Autoleucel Injection;
17. Patients previously received CAR-T cell therapy.
18. Other circumstances where the researcher deems it inappropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-27 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | Up to 28 days post-infusion
  Therapy-related adverse events (AE), including severe adverse events (SAE) and laboratory outliers with clinical significance, will be recorded and assessed according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
The safe dosage for a single infusion of Inaticabtagene Autoleucel Injection | Up to 28 days post-infusion
  The safe dosage for AIHA patients will be evaluated by comprehensively assessing the Overall Response Rate (ORR) and the incidence of adverse events (AEs).

SECONDARY OUTCOMES:
Overall Remission Rate (ORR) | Sixs months after cell reinfusion
  The proportion of subjects achieving CR, CRi or PR after treatment by Inaticabtagene Autoleucel Injection. CR is defined as clinical symptoms disappear, Hb≥110g/L (female) or Hb≥120g/L (male); the levels of hemolysis-related laboratory indicators (serum bilirubin and lactate dehydrogenase) return to normal. For CAD patients, CR criteria also include: undetectable clonal B cells and clonal IgM. Hematological complete remission with compensatory hemolytic state (CRi) is defined as Hb≥110g/L (female) or Hb≥120g/L (male); and hemolysis-related laboratory indicators (serum bilirubin and lactate dehydrogenase) improve but do not return to normal levels. Partial response (PR) is defined as Hb ≥ 100 g/L or an increase of ≥ 20 g/L from baseline; and at least 7 days without blood transfusion.
Changes in laboratory test indicators | Up to 24 months post-infusion
  Changes in Hemoglobin,reticulocytes, serum bilirubin, lactate dehydrogenase, and haptoglobin; clonal B cells and monoclonal immunoglobulin.
Drug-free Remission (DFR) | Up to 24 months post-infusion
  The duration from achieving CR, CRi, or PR to the time of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China

IPD SHARING:
Plan to Share IPD: No